CLINICAL TRIAL: NCT00860028
Title: Varenicline for Smoking Cessation in Heavy Drinking Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAA-O'Malley-P50AA15632-2009; P50AA015632 (NIH)
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Nicotine Dependence; Smoking; Heavy Drinking
Keywords: Smoking cessation; Smoking; Tobacco; Varenicline; Alcohol
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended Varenicline Pretreatment (Experimental): Arm 1 (Experimental) = 4 weeks varenicline (Chantix) titrated to 1 mg oral tablet twice per day before the smoking quit date followed by 4 weeks varenicline (Chantix) 1 mg oral tablet twice per day treatment.
  Interventions: Drug: Extended Varenicline Pretreatment
- Short-term Varenicline Pretreatment (Experimental): Arm 2 (Experimental) = 3 weeks placebo + 1 week varenicline (Chantix)pretreatment + 4 weeks varenicline 1 mg oral tablet twice per day treatment following the smoking quit date.
  Interventions: Drug: Short-term Varenicline Pretreatment

INTERVENTIONS:
Drug: Extended Varenicline Pretreatment — 4 weeks varenicline (Chantix) titrated to 1 mg oral tablet twice per day before the smoking quit date followed by 4 weeks varenicline (Chantix) 1 mg oral tablet twice per day treatment.
  Other Names: chantix
  Arms: Extended Varenicline Pretreatment
Drug: Short-term Varenicline Pretreatment — 3 weeks placebo + 1 week varenicline (Chantix)pretreatment + 4 weeks varenicline 1 mg oral tablet twice per day treatment following the smoking quit date.
  Other Names: Placebo
  Arms: Short-term Varenicline Pretreatment

SUMMARY:
The purpose of this study is to determine whether extended pretreatment with varenicline (Chantix) is more efficacious for smoking cessation than standard pretreatment, how well varenicline is tolerated in heavy drinking smokers, and whether varenicline reduces alcohol consumption.

DETAILED DESCRIPTION:
Smoking rates are elevated among drinkers compared to non-drinkers (Marks et al., 1997). Moreover, there is some evidence that both smokers who drink alcohol are less successful quitting smoking (Leeman, Huffman, & O'Malley, 2007). Thus, identifying interventions that are effective in reducing both smoking and heavy drinking in this population is warranted. Varenicline, a medication recently approved by the FDA, results in smoking cessation rates as high as 50%, significantly better than bupropion or placebo. There is preliminary experimental evidence from both animal and human laboratory research that varenicline reduces alcohol seeking and consumption (McKee, 2008; Steensland et al., 2007).

The typical dose schedule for varenicline involves a 1 week pretreatment phase prior to quitting smoking (Gonzales et al., 2006; Jorenby et al., 2006; Nides et al., 2006). However, greater quit rates have been observed 1 month after using varenicline compared to 1 week. Therefore, it is possible that extended pretreatment with varenicline may also yield better cessation outcomes than the standard 1 week lead in period. This may be particularly true if pretreatment also reduces alcohol consumption prior to the quit attempt.

Thirty regular smokers who drink alcohol heavily will receive open-label varenicline for 5 weeks according to the recommended titration schedule up to 1mg varenicline twice daily. Prior to the smoking quit date, subjects will be randomized to receive either extended pretreatment with varenicline (titration up to 1mg) for 4 weeks or short-term varenicline pretreatment (3 weeks placebo followed by 1 week of varenicline).

The primary aims of the study are to examine: (a) the efficacy of extended varenicline pretreatment for smoking cessation, (b) the safety and tolerability of varenicline in heavy drinking smokers, and (c) the efficacy of varenicline for reducing alcohol consumption in human participants. Effect size estimates for prolonged smoking abstinence and heavy drinking will be generated for a NIH grant application.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 75.
2. Smoking 5 or more cigarettes per occasion at least 3 times per week.
3. Fewer than 3 months of smoking abstinence in the past year.
4. Motivated to stop smoking.
5. Report exceeding maximum weekly drinking limits every week in the past 4 weeks and exceeding maximum daily drinking limits on at least 1 occasion in the past 4 weeks. Weekly heavy drinking is defined as 8 or more drinks for women and 15 or more drinks for men. Daily heavy drinking is defined as 4 or more drinks for women and 5 or more drinks for men on an occasion.

Exclusion Criteria:

1. Exhibit current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation
2. Any unexplained elevations in liver enzymes (i.e., transaminases, bilirubin)
3. Clinically significant cardiovascular disease
4. Uncontrolled hypertension
5. Hepatic or renal impairment
6. Severe chronic obstructive pulmonary disease
7. Diabetes mellitus requiring insulin or oral hypoglycemic medications.
8. Baseline systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 95 mm Hg
9. History of cancer (except treated basal cell or squamous cell carcinoma of the skin).
10. History of clinically significant allergic reactions.
11. Exhibit serious psychiatric illness (i.e., schizophrenia, bipolar disorder, severe major depression, panic disorder, borderline personality disorder, organic mood or mental disorders, or substantial suicide or violence risk) by history or psychological examination)
12. Have a current diagnosis of DSM-IV drug dependence other than nicotine or alcohol.
13. Have a current Diagnostic and Statistical Manual Diploma in Social Medicine IV (DSM-IV) diagnosis of alcohol dependence that is clinically severe defined by a) a history of seizures, delirium, or hallucinations during alcohol withdrawal, b) a Clinical Institute Withdrawal Assessment scale (Sullivan et al., 1989) score of > 8, c) report drinking to avoid withdrawal symptoms, or d) have had prior treatment of withdrawal.
14. Use of another investigational drug within 30 days.
15. Intention to donate blood or blood products during the treatment phase of the study.
16. Use of tobacco products other than cigarettes or use of marijuana.
17. Use of nicotine replacement therapy, clonidine, varenicline, bupropion, or nortriptyline within the month prior to enrollment or intention to use medication that might interfere with study medication.
18. Body Mass Index (calculated as weight in kilograms divided by the square of height in meters) less than 15 or greater than 38 or weight less than 45 kg.
19. Females of childbearing potential who are pregnant, nursing, or not practicing effective contraception (oral, injectable, or implantable contraceptives, intrauterine device, or barrier method with spermicide).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie S O'Malley, PhD, Principal Investigator — Yale University

REFERENCES:
- [Result] Fucito LM, Toll BA, Wu R, Romano DM, Tek E, O'Malley SS. A preliminary investigation of varenicline for heavy drinking smokers. Psychopharmacology (Berl). 2011 Jun;215(4):655-63. doi: 10.1007/s00213-010-2160-9. Epub 2011 Jan 11. PMID 21221531
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient research clinic
Pre-assignment Details: Prior to randomization, inclusion and exclusion criteria were assessed. Reasons for exclusion included health problems, not meeting drinking/smoking criteria, other drug use, and depression requiring treatment.
Groups:
- Extended Varenicline Pretreatment: Arm 1 (Experimental) = 3 weeks varenicline (Chantix) 1 mg oral tablet twice per day pretreatment + 5 weeks varenicline (Chantix) 1 mg oral tablet twice per day treatment.
Period: Placebo Controlled Pretreatment Period
Arm/Group | Extended Varenicline Pretreatment | Short-term Varenicline Pretreatment
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1
Not completed — No longer interested in treatment | 2 | 1
Period: Smoking Cessation Phase
Arm/Group | Extended Varenicline Pretreatment | Short-term Varenicline Pretreatment
Started | 13 | 14
Completed | 13 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Short Varenicline Pretreatment (Placebo): Arm 2 (Experimental) = 3 weeks placebo pretreatment + 5 weeks varenicline (Chantix) 1 mg oral tablet twice per day treatment
- Total: Total of all reporting groups
Arm/Group | Extended Varenicline Pretreatment | Short Varenicline Pretreatment (Placebo) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.87 (8.52) | 43.47 (7.99) | 43.17 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Continuous Smoking Abstinence in the Extended Varenicline Pretreatment Versus Short-term Varenicline Pretreatment Conditions.
Description: Compares the number of participants who reported no smoking, not even a puff, from the quit date through until the end of treatment (i.e., last 4 weeks of treatment) in the varenicline versus placebo pretreatment conditions.
Time Frame: Last 4 weeks of treatment
Population: All participants were included in the analysis, assuming an intention to treat method.
Measure: Number; unit: Participants
Groups:
- Extended Varenicline Pretreatment: Arm 1 (Experimental) = 4 weeks varenicline (Chantix) titrated to 1 mg oral tablet twice per day pretreatment + 4 weeks varenicline (Chantix) 1 mg oral tablet twice per day treatment following the smoking quit date
Arm/Group | Extended Varenicline Pretreatment | Short-term Varenicline Pretreatment
Number analyzed (Participants) | 15 | 15
Participants | 4 | 2
Statistical Analysis 1: Comparison: Extended Varenicline Pretreatment vs Short-term Varenicline Pretreatment; Test type: Superiority or Other; p = 0.36, Chi-squared

2. Primary Outcome: Mean Percentage of Heavy Drinking Days Comparing Participants in the Extended Varenicline Pretreatment Versus Short-term Varenicline Pretreatment Conditions
Description: Compares the mean percentage of heavy drinking days over the 3-week placebo-controlled pretreatment phase comparing participants in the extended varenicline pretreatment versus the short-term varenicline pretreatment conditions. Heavy drinking defined as consuming 4 or more drinks per occasion for women and 5 or more drinks per occasion for men. Drinking in the final week of pretreatment prior to the quit-date is not included because both groups were receiving active varenicline during this period.
Time Frame: First 3 weeks (pretreatment)
Population: All participants were included in the analysis, assuming an intention to treat method.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Extended Varenicline Pretreatment | Short-term Varenicline Pretreatment
Number analyzed (Participants) | 15 | 15
percentage of heavy drinking days | 22.7 (17.5) | 38.0 (31.2)
Statistical Analysis 1: Comparison: Extended Varenicline Pretreatment vs Short-term Varenicline Pretreatment; Test type: Superiority or Other; p = 0.06, General Linear Model

3. Secondary Outcome: Number of Participants Who Reported an Adverse Event in the Varenicline Pretreatment Versus Placebo Pretreatment Conditions
Description: Compares the number of participants who reported an adverse event in the extended varenicline pretreatment versus short-term varenicline pretreatment conditions during the 3-week placebo controlled pretreatment phase
Time Frame: First 3 weeks (pretreatment)
Population: All participants were included in the analysis, assuming an intention to treat method.
Measure: Number; unit: Number of participants
Arm/Group | Extended Varenicline Pretreatment | Short-term Varenicline Pretreatment
Number analyzed (Participants) | 15 | 15
Number of participants | 10 | 3
Statistical Analysis 1: Comparison: Extended Varenicline Pretreatment vs Short-term Varenicline Pretreatment; Test type: Superiority or Other; p = 0.03, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events also assessed post quitting smoking during the open label phase of the study.
Arm/Group | Extended Varenicline Pretreatment | Short Varenicline Pretreatment (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Varenicline Pretreatment (N=15) | Short Varenicline Pretreatment (Placebo) (N=15)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) — Report of moderate constipation greater than baseline ratings.
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 7 (7)
Acid Reflux (Gastrointestinal disorders) | 4 (4) | 7 (7)
Anxiety (Psychiatric disorders) | 4 (4) | 4 (4)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Decreased Appetite (General disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Dry Mouth (General disorders) | 4 (4) | 4 (4)
Dysgeusia (General disorders) | 4 (4) | 7 (7)
Edema (Vascular disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 8 (8) | 6 (6)
Flatulence (Gastrointestinal disorders) | 6 (6) | 6 (6)
Headache (General disorders) | 5 (5) | 8 (8)
Increased Appetite (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Increased Bowel (Gastrointestinal disorders) | 2 (2) | 5 (5)
Indigestion (Gastrointestinal disorders) | 6 (6) | 3 (3)
Insomnia (General disorders) | 7 (7) | 8 (8)
Itching (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Labored Breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lethargy (General disorders) | 5 (5) | 5 (5)
Missed Period (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 7 (7)
Nightmares (General disorders) | 2 (2) | 1 (1)
Nose Mucus (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Sleepiness (General disorders) | 6 (6) | 3 (3)
Sweating (Endocrine disorders) | 4 (4) | 7 (7)
Upper Respiratory Problem (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Vivid Dreams (General disorders) | 10 (10) | 12 (12)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Other (General disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No